CLINICAL TRIAL: NCT05560269
Title: Comparing Verbal Cueing and the Constraint-Led Approach for Teaching the Kettlebell Swing
Brief Title: Verbal Cueing vs Constraint-Led Approach for Teaching the Kettlebell Swing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004623
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Movement Disorders; Muscle Tenderness
MeSH Terms: conditions — Movement Disorders; Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- verbal and physical constraint group (Experimental): Use of verbal and physical constraint
  Interventions: Behavioral: Verbal coaching vs. Constraint based coaching
- verbal constraint group (Active Comparator): Use of verbal constraint only
  Interventions: Behavioral: Verbal coaching vs. Constraint based coaching
- physical constraint group (Experimental): Use of constraint only
  Interventions: Behavioral: Verbal coaching vs. Constraint based coaching

INTERVENTIONS:
Behavioral: Verbal coaching vs. Constraint based coaching — * 15 repetitions of kettlebell swings using verbal cues and physical constraints to teach the second part of the movement → 30 seconds to 1 minute rest interval→ 15 repetitions of kettlebell swings using verbal cues and physical constraints to combine both parts of the movement → 30 seconds to 1 minute rest interval
  * 15 repetitions of kettlebell swings using verbal cues to teach the second part of the movement → 30 seconds to 1 minute rest interval→ 15 repetitions of kettlebell swings using verbal cues to combine both parts of the movement → 30 seconds to 1 minute rest interval
  * 15 repetitions of kettlebell swings using physical constraints to teach the second part of the movement → 30 seconds to 1 minute rest interval→ 15 repetitions of kettlebell swings using physical constraints to combine both parts of the movement → 30 seconds to 1 minute rest interval

SUMMARY:
The purpose of this study is to determine which method is most effective for teaching the kettlebell swing: verbal cueing, physical constraints, or a combination of the two.

DETAILED DESCRIPTION:
There is a method of teaching and learning movement and exercise skills known as the constraint-led approach. This method of movement learning has the learner exploring and experimenting different variations of an exercise by self-organizing around a set of given constraints of the individual, environment and task. Individual constraints are qualities about the person performing the task such as their arm length and height. Environmental constraints regard the environment where the task is being performed and include factors such as lighting and temperature. Finally, the task constraints are qualities about the movement and exercises being performed such as asking someone to do a half squat onto a box instead of a full bodyweight squat in the air. This constraints way of teaching movement has the movement educator as a guide or architect that shapes the qualities of the task the learner must navigate.

The kettlebell swing was chosen as the primary exercise for this study due to its efficacy and practicality as a functional movement pattern. Current literature suggests that kettlebell swings may elicit an increase in strength measured in the form of a deadlift exercise, which may have carry over to activities of daily living, such as bending over to lift a box with proper form. In a 2016 study, Edinborough et al. examined the proposed implications that repeated kettlebell swings could be used as a practical tool to increase endurance capacity of the lumbar extensor complex. The investigators of this study found that after a 60 second bout of continuous kettlebell swings, participants demonstrated a reduction in isometric strength, demonstrating fatigue of this musculature. The implications of this study suggest that kettlebell swings may increase the fatigue threshold of the lumbar extensor musculature, which may provide protective measures regarding the development of musculoskeletal conditions such as low back pain, as a decrease in activation of these associated muscles may be apparent during periods of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 55 years.
* Subjective rating of 3/5 or less on confidence with kettlebell swings.

Exclusion Criteria:

* Inability to read and write in English.
* Previous injury to the lower extremity that prevents normal squatting motion.
* Physical Activity Readiness Questionnaire suggesting inability to safely participate in exercise.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Hip range of motion | Base line and immediately after intervention
  Joint angles of the subject's dominant side of the hip will be measured from a horizontal view using the OnForm app on the ipad. Subjects will have yellow, circular stickers placed on bony landmarks such as the greater trochanter, lateral femoral epicondyle, lateral malleolus, and the tuberosity of the 5th metatarsal. The participant will be performing the kettlebell swings without shoes for standardization purposes. These measurements will be compared both pre- and post-test to measure any changes.
Knee range of motion | Base line and immediately after intervention
  Joint angles of the subject's dominant side of the knee will be measured from a horizontal view using the OnForm app on the ipad (as shown below). Subjects will have yellow, circular stickers placed on bony landmarks such as the greater trochanter, lateral femoral epicondyle, lateral malleolus, and the tuberosity of the 5th metatarsal. The participant will be performing the kettlebell swings without shoes for standardization purposes. These measurements will be compared both pre- and post-test to measure any changes.
Ankle range of motion | Base line and immediately after intervention
  Joint angles of the subject's dominant side of the ankle will be measured from a horizontal view using the OnForm app on the ipad (as shown below). Subjects will have yellow, circular stickers placed on bony landmarks such as the greater trochanter, lateral femoral epicondyle, lateral malleolus, and the tuberosity of the 5th metatarsal. The participant will be performing the kettlebell swings without shoes for standardization purposes. These measurements will be compared both pre- and post-test to measure any changes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine NA, Hasan MB, Avalos MA, Lee S, Rigby BR, Kwon YH. Effects of kettlebell mass on lower-body joint kinetics during a kettlebell swing exercise. Sports Biomech. 2022 Oct;21(9):1032-1045. doi: 10.1080/14763141.2020.1726442. Epub 2020 Mar 4. PMID 32131695
- [Background] McGill SM, Marshall LW. Kettlebell swing, snatch, and bottoms-up carry: back and hip muscle activation, motion, and low back loads. J Strength Cond Res. 2012 Jan;26(1):16-27. doi: 10.1519/JSC.0b013e31823a4063. PMID 21997449
- [Background] Lyons BC, Mayo JJ, Tucker WS, Wax B, Hendrix RC. Electromyographical Comparison of Muscle Activation Patterns Across Three Commonly Performed Kettlebell Exercises. J Strength Cond Res. 2017 Sep;31(9):2363-2370. doi: 10.1519/JSC.0000000000001771. PMID 28394829
- [Background] Andersen V, Fimland MS, Gunnarskog A, Jungard GA, Slattland RA, Vraalsen OF, Saeterbakken AH. Core Muscle Activation in One-Armed and Two-Armed Kettlebell Swing. J Strength Cond Res. 2016 May;30(5):1196-204. doi: 10.1519/JSC.0000000000001240. PMID 26473519
- [Background] Otte FW, Rothwell M, Woods C, Davids K. Specialist Coaching Integrated into a Department of Methodology in Team Sports Organisations. Sports Med Open. 2020 Nov 16;6(1):55. doi: 10.1186/s40798-020-00284-5. PMID 33196910